CLINICAL TRIAL: NCT03604016
Title: Pilot Study to Assess the Antiviral Activity and Safety of Besifovir Dipivoxil 150mg and L-carnitine 660mg Compared to Tenofovir Alafenamide 25mg in Chronic Hepatitis B Patients With Nonalcoholic Fatty Liver
Brief Title: Study to Assess Efficacy of Besifovir and L-carnitine in Chronic Hepatitis B Patients With Nonalcoholic Fatty Liver
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID-BVCL-401
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Carnitine; tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Besifovir dipivoxil+L-carnitine (Experimental): Besifovir dipivoxil 150 mg and L-carnitine 330 mg
  Interventions: Drug: Besifovir dipivoxil; Drug: L-carnitine
- Tenofovir Alafenamide (Active Comparator): Tenofovir Alafenamide 25mg
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Besifovir dipivoxil — Besifovir dipivoxil 150 mg
  Arms: Besifovir dipivoxil+L-carnitine
Drug: L-carnitine — Besifovir dipivoxil 150 mg
  Arms: Besifovir dipivoxil+L-carnitine
Drug: Tenofovir Alafenamide — Tenofovir Alafenamide 25mg
  Arms: Tenofovir Alafenamide

SUMMARY:
Pilot study to assess the antiviral activity and safety of Besifovir dipivoxil 150mg and L-carnitine 660mg compared to Tenofovir Alafenamide 25mg in chronic hepatitis B patients with Nonalcoholic fatty liver

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age and older, Male or female patients
* Chronic hepatitis B patients with Nonalcoholic fatty liver
* Patients who use oral anti-diabetic drug or drugs for hyperlipemia without any change in drug dosage within 2 month before screening visit
* Patients who have been explained about the trial and agreed to the consent
* Patients who agree with the approved method of contraception during the clinical trial

Exclusion Criteria:

* Patients with hepatitis C virus, hepatitis D virus or human immunodeficiency virus
* Patients who has a history of liver transplantation or Child-Pugh score >=8
* Alpha-fetoprotein (AFP) > 50 ng/mL or Hepatocellular Carcinoma (HCC) patients
* Patients who have taken Besifovir or Vemlidy
* Among the patients treated with immunosuppressive drug within 6 months before screening, suspected case of the declined immunity in the opinion of the investigator
* Chronic alcoholism (Significant alcohol consumption: male > 210 g/week, female> 140 g/week)
* Patients who take drugs that can cause hepatic steatosis
* Patient diagnosed with a malignant tumor within 5 years before screening or relapsed patient
* Patients with uncontrolled diabetes mellitus (HbA1c > 9%) or using insulin
* Patients who participate in other clinical trials or is supposed to do so during the study period
* Pregnant or breast-feeding women or women who have plan to be pregnant.
* Patients with a history of hypersensitivity to the test drug or the components of the test drug
* Patients with moderate or severe renal impairment
* Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* History within the past one years or presence of drug abuse or alcoholism.
* Patient has serious disease judged by investigator such as heart failure, renal failure, and pancreatitis
* Patient has liver diseases except chronic hepatitis B (i.e. hematochromatosis, alcoholic liver disease, nonalcoholic fatty liver disease, alpha-1 antitrypsin deficiency etc.)
* Patient has history of organ transplantation
* Patient concerned about the decline in daily activity or not able to understand the objectives and methods due to the psychiatric problems
* Patients who are considered to be unacceptable in this study under the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-09-23 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 116 copies/mL (20 IU/mL)) at the 48 week | at the 48th week

SECONDARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 116 copies/mL (20 IU/mL)) at the 24 week | at the 24th week

OTHER OUTCOMES:
The change of liver fat at 48 weeks | at the 48th weeks